CLINICAL TRIAL: NCT01532908
Title: A Phase II Open-Label Study of the Clinical Effectiveness of a Human Monoclonal Antibody Against Hepatitis C Virus E2 Glycoprotein (MBL-HCV1) Combined With Oral Direct-Acting Antivirals in Hepatitis C Infected Patients Undergoing Liver Transplantation
Brief Title: Open Label Study of the Efficacy and Safety of MBL-HCV1 in Combination With Oral Direct-Acting Antivirals in Patients Undergoing Liver Transplantation for Hepatitis C
Acronym: MBL-HCV1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to funding constraints
Sponsor: MassBiologics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MBL-HCV1-11-03
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis C Infection
Keywords: Liver Transplantation
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: MBL-HCV1 and Telaprevir (Experimental)
  Interventions: Biological: MBL-HCV1; Drug: Telaprevir (Part 1)
- Part 2: MBL-HCV1 and Sofosbuvir (Experimental)
  Interventions: Biological: MBL-HCV1; Drug: Sofosbuvir (Part 2)

INTERVENTIONS:
Biological: MBL-HCV1 — 50 mg/kg MBL-HCV1, intravenous, up to 15 infusions over 56 days; option for extended treatment through 84 days if viral load undetectable at day 56
Drug: Telaprevir (Part 1) — Two 375 mg tablets, 3 times a day up to 56 days; option for extended treatment through 84 days if viral load undetectable at day 56
  Other Names: Incivek (telaprevir)
  Arms: Part 1: MBL-HCV1 and Telaprevir
Drug: Sofosbuvir (Part 2) — One 400 mg tablet, 1 time per day up to 56 days; option for extended treatment through 84 days if viral load undetectable at day 56
  Other Names: Sovaldi (sofosbuvir)
  Arms: Part 2: MBL-HCV1 and Sofosbuvir

SUMMARY:
The purpose of this study is to assess efficacy of a human monoclonal antibody against Hepatitis C (MBL-HCV1) combined with telaprevir [part 1: an HCV protease inhibitor] or sofosbuvir [part 2: an Hepatitis C virus NS5B polymerase inhibitor] in a 56 day treatment duration in patients undergoing liver transplantation due to chronic HCV infection. There is an option for extended study treatment through 84 days if viral load is undetectable at day 56.

DETAILED DESCRIPTION:
Administration of Intravenous infusions of MBL-HCV1 (50mg/kg) human monoclonal antibody during the first 14 days post-transplantation: three infusions on day 0 (1-4 hours prior to the anhepatic phase, during the anhepatic phase, and 4-12 hours post-reperfusion). Daily infusions on days 1 through 7, weekly infusions on day 14 ± 2, day 21 ± 3, and day 28 ± 3, followed by biweekly infusions on day 42 ± 3 and on day 56 ± 3 if criteria for the stopping rule are not met. For those subjects electing extended treatment, the administration of additional infusions on day 70 ± 3 and day 84 ± 3 will be performed. Subjects receive an oral direct-acting antiviral (telaprevir in Part 1 and sofosbuvir in Part 2) starting no earlier than day 3 post-transplant and no later than day 7; dosing continuing through day 56 unless criteria for the stopping rule are met. Subjects who elect to receive extended study treatment for a total of 12 weeks continue telaprevir in Part 1 or sofosbuvir in Part 2 through day 84 ± 3.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age with documented chronic hepatitis C virus infection of genotype 1 undergoing liver transplantation from either a deceased donor or living donor.
* Patient or legal guardian/health care proxy must have read, understood and provided written informed consent and HIPAA authorization after the nature of the study has been fully explained.

Exclusion Criteria:

* Positive for hepatitis B surface Antigen
* Positive serology for HIV
* Pregnancy or Breastfeeding
* Previous history of any organ transplant
* Planned receipt of combined organ transplant (e.g. liver and kidney)
* Receipt or planned receipt of immune globulin (IVIG) within 90 days of enrollment
* Extrahepatic malignancy not currently in remission and/or receiving systemic chemotherapy and/or radiation within 90 days prior to enrollment. Exceptions include chemoembolization for hepatocellular carcinoma or cutaneous malignancies managed with local treatment
* Hepatocellular carcinoma with tumor burden outside of the Milan criteria
* Serum creatinine > 2.5 for > or = six months at the time of enrollment
* Personal or family history (first degree relative) of deep venous thrombosis or pulmonary embolism
* Receipt of liver allograft from HCV positive donor or Hepatitis B core antibody positive donor
* Receipt of liver allograft donated after cardiac death of donor
* Receipt of any antiviral agents (licensed or investigational) for hepatitis C virus within 30 days prior to liver transplantation, unless patient has documented detectable HCV RNA during this 30 day period
* Previous receipt of an HCV protease inhibitor (for subjects enrolling in Part 1: telaprevir)
* Receipt of any other investigational study product within 30 days prior to enrollment
* Seizure disorder requiring anti-convulsant therapy
* Pulmonary arterial hypertension requiring sildenafil or tadalafil infusion (for subjects enrolling in Part 1: telaprevir)
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the patient participating in the study or make it unlikely that the patient could complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas

REFERENCES:
- [Background] Smith HL, Chung RT, Mantry P, Chapman W, Curry MP, Schiano TD, Boucher E, Cheslock P, Wang Y, Molrine DC. Prevention of allograft HCV recurrence with peri-transplant human monoclonal antibody MBL-HCV1 combined with a single oral direct-acting antiviral: A proof-of-concept study. J Viral Hepat. 2017 Mar;24(3):197-206. doi: 10.1111/jvh.12632. Epub 2016 Nov 7. PMID 28127942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chronically infected patients with HCV genotype 1a (Part 1) or genotype 1 (Part 2) scheduled to undergo a liver transplantation were recruited at 5 U.S. transplantation centers between May 2012 and August 2015. Eleven subjects were enrolled. Ten subjects were transplanted and received study intervention in the study (8 in Part 1) and (2 in Part 2).
Pre-assignment Details: Reasons for exclusion from study treatment included receipt of an ineligible organ at time of transplant, awaiting transplant at time study enrollment stopped, became ineligible, withdrew consent and subject expired prior to organ offer.
Period: Overall Study
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir
Started | 9 | 2
Infused | 9 | 2
Transplanted | 8 | 2
Completed | 8 | 2
Not Completed | 1 | 0
Not completed — Not Transplanted | 1 | 0

BASELINE CHARACTERISTICS:
Population: The ten subjects (8 in Part 1 and 2 in Part 2) who initiated study infusions, underwent liver transplantation and received an oral direct-acting antiviral (telaprevir in Part 1 or sofosbuvir in Part 2) were included in the analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Continuous [Mean (Full Range); unit: years] | 59 [53 to 63] | 56 [56 to 56] | 58 [53 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Hepatocellular Carcinoma [Count of Participants; unit: Participants] — The number of participants with a history of hepatocellular carcinoma prior to liver transplantation was reported
  Participants | 7 | 1 | 8
Baseline serum HCV RNA concentration [Mean (Full Range); unit: Log10 IU/mL] — Participants' pre-transplant baseline serum HCV RNA concentration was measured by quantitative RT-PCR (reverse-transcriptase PCR)
  Log10 IU/mL | 5.53 [4.02 to 6.49] | 6.25 [6.15 to 6.34] | 5.67 [4.02 to 6.49]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Undetectable HCV RNA at Day 56 Post Liver Transplantation
Description: The primary outcome was to determine if MBL-HCV1 in combination with the oral direct-acting antiviral could reduce HCV viral RNA to undetectable at day 56 post transplant and prevent the new liver from becoming productively infected. Undetectable HCV RNA was defined as the level below the lower limit of detection (LLOD) of an FDA-approved polymerase chain reaction (PCR) assay. HCV RNA was quantified by PCR (e.g., COBAS®AmpliPrep/ COBAS® TaqMan® HCV Test manufactured by Roche or equivalent) at each study site
Time Frame: Day 56
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir
Number analyzed (Participants) | 8 | 2
Participants | 4 | 2

2. Secondary Outcome: Safety and Tolerability of Study Treatment by Number of Adverse Events Reported
Description: Adverse events were assessed by targeted medical history, physical examinations and laboratory testing. Abnormal laboratory values constituted adverse events only if they induced clinical signs or symptoms and/or required therapy that was new or enhanced from baseline. Solicited adverse reactions included the occurrence of the following during or immediately after the infusion: arthralgia, chills, dyspnea, fatigue, fever, headache, nausea, hives, or rash. The presence of any of these symptoms (new or worsening from baseline) was documented as an adverse event. In addition, subjects were asked at all scheduled study visits to report any other adverse events. Adverse events were summarized by System Organ Class (SOC) using MedDRA (version 14.1)
Time Frame: Day 0 start of first infusion through Day 56 or six weeks after last dose of study treatment whichever is later, up to approximately 126 days
Population: as for baseline characteristics
Measure: Number; unit: Events
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir
Number analyzed (Participants) | 8 | 2
Events
  Blood And Lymphatic System Disorders | 6 | 0
  Cardiac Disorders | 0 | 1
  Eye Disorders | 1 | 0
  Gastrointestinal Disorders | 9 | 3
  General Disorders And Administration Site Conditions | 12 | 0
  Hepatobiliary Disorders | 3 | 0
  Immune System Disorders | 2 | 1
  Infections And Infestations | 6 | 2
  Injury, Poisoning And Procedural Complications | 11 | 1
  Investigations | 3 | 1
  Metabolism And Nutrition Disorders | 14 | 2
  Musculoskeletal And Connective Tissue Disorders | 1 | 1
  Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) | 0 | 1
  Nervous System Disorders | 6 | 1
  Psychiatric Disorders | 5 | 2
  Renal And Urinary Disorders | 1 | 0
  Reproductive System And Breast Disorders | 1 | 2
  Respiratory, Thoracic And Mediastinal Disorders | 10 | 0
  Skin And Subcutaneous Tissue Disorders | 2 | 1
  Surgical And Medical Procedures | 0 | 1
  Vascular Disorders | 5 | 1

3. Secondary Outcome: Number of Subjects With Undetectable Serum HCV RNA at Study Day 7, 10, 14, 28, 35, 42, 49, 70, 84 and 98 in Liver Transplant Recipients and for Those Subjects Receiving an Additional 4 Weeks of Treatment at Study Day 105, 112 and 126
Description: The number of subjects with undetectable HCV RNA by study visit day was analyzed utilizing a "last value carried forward" (LVCF) strategy so that each study visit day had data from (8 subjects in Part 1 and 2 subjects in Part 2), effectively imputing the information for the subjects who had missing data due to a missed study visit, HCV RNA measured with a non-FDA approved assay, or completion of all required post-treatment study visits. The last recorded HCV RNA status for a subject (detectable vs undetectable) was used for the next missing level (in ascending visit number order) until a new HCV RNA level was recorded at a later visit. Serum HCV RNA was measured by Quantitative RT-PCR using an FDA-approved quantitative assay
Time Frame: Day 7, 10, 14, 28, 35, 42, 49, 70, 84, 98, 105, 112 and 126
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir
Number analyzed (Participants) | 8 | 2
participants
  Day 7 | 0 | 0
  Day 10 | 2 | 0
  Day 14 | 2 | 0
  Day 28 | 4 | 2
  Day 35 | 5 | 2
  Day 42 | 5 | 2
  Day 49 | 5 | 2
  Day 70: number analyzed (Participants) | 3 | 2
  Day 70 | 3 | 2
  Day 84: number analyzed (Participants) | 3 | 2
  Day 84 | 2 | 2
  Day 98: number analyzed (Participants) | 3 | 2
  Day 98 | 2 | 2
  Day 105: number analyzed (Participants) | 3 | 2
  Day 105 | 2 | 2
  Day 112: number analyzed (Participants) | 3 | 2
  Day 112 | 2 | 2
  Day 126: number analyzed (Participants) | 3 | 2
  Day 126 | 2 | 2

4. Secondary Outcome: Change in Viral Load Between Baseline Pre-transplant HCV RNA Levels and Study Day 7, 10, 14, 28, 35, 42, 49, 56, 70, 84 and 98 in Liver Transplant Recipients
Description: Serum HCV RNA was measured by quantitative RT-PCR. The change in log 10 IU/mL HCV viral load from baseline was compared with pre-transplant HCV RNA level and evaluated for each subject at each study visit.
  Change in the level of HCV RNA in serum, log10(IU/mL), is defined as the difference between the level measured at Baseline and the specified time point. If HCV RNA was not detected by the PCR assay, the lower level of detection of the PCR assay was used for the calculation
Time Frame: Baseline pre-transplant and study Day 7, 10, 14, 28, 35, 42, 49, 56, 70, 84 and 98
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: Log10 IU/mL
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir
Number analyzed (Participants) | 8 | 2
Log10 IU/mL
  Day 7 | -2.97 [-3.94 to -2.45] | -3.46 [-3.57 to -3.35]
  Day 10 | -3.35 [-4.32 to -2.20] | -3.99 [-4.38 to -3.60]
  Day 14 | -3.58 [-4.70 to -1.87] | -4.32 [-4.85 to -3.80]
  Day 28 | -2.94 [-5.54 to 1.57] | -5.29 [-5.38 to -5.19]
  Day 35 | -3.01 [-5.54 to 1.69] | -5.29 [-5.38 to -5.19]
  Day 42 | -2.94 [-5.54 to 1.80] | -5.29 [-5.38 to -5.19]
  Day 49 | -2.89 [-5.54 to 1.78] | -5.29 [-5.38 to -5.19]
  Day 56 | -2.28 [-5.54 to 1.86] | -5.29 [-5.38 to -5.19]
  Day 70 | -2.62 [-5.54 to 1.39] | -5.29 [-5.38 to -5.19]
  Day 84 | -2.53 [-5.16 to 1.41] | -5.29 [-5.38 to -5.19]
  Day 98 | -0.76 [-4.62 to 1.48] | -5.29 [-5.38 to -5.19]

5. Secondary Outcome: Number of Participants With HCV Resistance-associated Variants to MBL-HCV1 and Oral Direct-acting Antivirals Before and After Receipt of Study Treatment
Description: Conventional sequencing was performed on HCV RNA isolated from a subset of serum samples obtained at baseline, at the time of viral rebound, and at the end of study in subjects who did not achieve a sustained virologic response. The targets of both the MBL-HCV1 antibody (E1/E2 glycoprotein) and telaprevir (NS3) were sequenced. The data displays the number of subjects with > 20% resistance associated variants (RAV) reported for the target MBL-HCV1 and/or Direct-acting Antiviral (DAA)
Time Frame: Pre-transplant, time of viral rebound (assessed from Day 7-Day 56 of treatment), end of study (up to day 126) in subjects who did not achieve a sustained virologic response (SVR)
Population: as for baseline characteristics
Measure: Number; unit: Participants with > 20 % RAV
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir
Number analyzed (Participants) | 8 | 2
Participants with > 20 % RAV
  Pre-transplant | 4 | NA — 1 For the Part 2: MBL-HCV1 and Sofosbuvir" Arm/Group Pre-transplant timepoint, virus was available but not analyzed because there was no viral rebound, therefore there was no virus available for comparison.
  Viral Rebound | 4 | NA — 2 For the Part 2: MBL-HCV1 and Sofosbuvir" Arm/Group both subjects had undetectable HCV RNA by day 21 and remained undetectable for 24 weeks post-treatment (SVR24), therefore there was no virus available for analysis.
  End of Study | 7 | NA — 2 For the Part 2: MBL-HCV1 and Sofosbuvir" Arm/Group both subjects had undetectable HCV RNA by day 21 and remained undetectable for 24 weeks post-treatment (SVR24), therefore there was no virus available for analysis.

6. Other Pre Specified Outcome: Number of Subjects With Sustained Virologic Response (SVR) at Week 12 and Week 24
Description: Number of subjects with sustained virologic response (defined as HCV RNA concentration below the limit of detection) at 12 and 24 weeks post-treatment was examined as an exploratory endpoint in subjects whose HCV RNA remained undetectable at the 6 week post-treatment safety follow-up visit.
  Those subjects that had detectable HCV RNA at the end of safety follow-up period were not assessed for SVR 12 and SVR 24. Those subjects achieving an SVR12 were assessed for the durability of the response at 24 weeks after the end of treatment
Time Frame: 12 weeks after the end of treatment (SVR12) and 24 weeks after the end of treatment 12 weeks and 24 weeks post-treatment
Population: Of 8 subjects in Part 1, 2 had undetectable HCV RNA at 6 wk post-treatment. Therefore, at wk 12 (day 168), per protocol, 2 were analyzed. 1 had detectable HCV RNA at wk 12. Per protocol, the subject did not require a 24 wk visit. The other subject had undetectable HCV RNA at wk 12. Therefore, only 1 subject was analyzed at wk 24 (day 252). This subject had undetectable HCV RNA at wk 24.
  2 subjects in Part 2 had undetectable HCV RNA at 12 & 24 wks. 2 subjects were analyzed at the 12 & 24 wks
Measure: Number; unit: participants
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir
Number analyzed (Participants) | 2 | 2
participants
  Post Treatment Week 12 | 1 | 2
  Post Treatment Week 24: number analyzed (Participants) | 1 | 2
  Post Treatment Week 24 | 1 | 2

ADVERSE EVENTS:
Time Frame: Day 0 start of first infusion through Day 56 or six weeks after last dose of study treatment whichever is later, up to approximately 126 days
Description: Adverse events were assessed by targeted medical history, physical examinations and laboratory testing. The following adverse reactions were solicited during or immediately after the infusion: arthralgia, chills, dyspnea, fatigue, fever, headache, nausea, hives, or rash. Summarized by System Organ Class (SOC) and Preferred Term (PT)
Arm/Group | Part 1: MBL-HCV1 and Telaprevir | Part 2: MBL-HCV1 and Sofosbuvir
Serious Adverse Events (participants affected / at risk) | 7/8 | 1/2
Other Adverse Events (participants affected / at risk) | 8/8 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MBL-HCV1 and Telaprevir (N=8) | Part 2: MBL-HCV1 and Sofosbuvir (N=2)
GENERALISED OEDEMA (General disorders) | 1 (1) | 0 (0) — AND ADMINISTRATION SITE CONDITIONS
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) — AND ADMINISTRATION SITE CONDITIONS
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
LIVER TRANSPLANT REJECTION (Immune system disorders) | 0 (0) | 1 (1)
TRANSPLANT REJECTION (Immune system disorders) | 2 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MBL-HCV1 and Telaprevir (N=8) | Part 2: MBL-HCV1 and Sofosbuvir (N=2)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GLOSSODYNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) — AND ADMINISTRATION SITE CONDITIONS
FATIGUE (General disorders) | 2 (2) | 0 (0) — AND ADMINISTRATION SITE CONDITIONS
OEDEMA (Gastrointestinal disorders) | 1 (1) | 0 (0) — AND ADMINISTRATION SITE CONDITIONS
OEDEMA PERIPHERAL (General disorders) | 3 (4) | 0 (0) — AND ADMINISTRATION SITE CONDITIONS
PYREXIA (General disorders) | 2 (2) | 0 (0) — AND ADMINISTRATION SITE CONDITIONS
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
INCISION SITE PRURITUS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 2 (2) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (3) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 1 (1)
VOCAL CORD PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (3) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
TESTICULAR SWELLING (Reproductive system and breast disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (3) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
REPERFUSION INJURY (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less